CLINICAL TRIAL: NCT02089022
Title: Analysis of Neuromuscular Responses and the Balance After the Application of Physiotherapy Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Thiago Batista Muniz, Master, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCRP 12788/2011
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Musculoskeletal Injuries; Cryotherapy Effect; Complication of Diathermy Procedure
Keywords: Ice; Heat; Ground reaction forces; Electromyography; Lower Limb; Center of pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physiotherapy resources (Experimental): The goal of applying ice and shortwave diathermy to the calf, ankle and sole of the foot was to verify the effect of this resources at the neuromuscular response of the lower limb and postural balance
  Interventions: Other: Physiotherapy resources

INTERVENTIONS:
Other: Physiotherapy resources — The application of ice has been accomplished by means of a plastic bag containing 1.5 kg of crushed ice. The duration of the application was 30 minutes. The use of shortwave diathermy was performed by means of rectangular electrodes having a duration of 20 minutes.

SUMMARY:
The aim of this study was to evaluate the effect of ice and shortwave diathermy in different regions of lower limb neuromuscular response and balance.

DETAILED DESCRIPTION:
Applying ice and shortwave diathermy was performed separately (on different days) in the foot, ankle and calf. To assess the neuromuscular response was evaluated electromyographic activity of the rectus femorals, biceps femorals, gastrocnemius and tibialis anterior. To assess the effect of applications on balance, through a force platform was evaluated oscillation of the center of pressure as well as ground reaction forces.

ELIGIBILITY:
Inclusion Criteria:

* woman
* healthy
* young
* sedentary

Exclusion Criteria:

* sensory changes
* history of fractures in the lower limbs
* being in the menstrual period
* diabetes Mellitus
* Bone, muscle and/or neural diseases

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Analysis of neuromuscular responses after the application of physiotherapy resources | We evaluated 22 volunteers in a period of one year and 6 months
  To evaluate the neuromuscular response, we used the median frequency of the electromyographic variables and root mean square
Analysis of body balance after the application of physiotherapy | We evaluated 22 volunteers in a period of one year and 6 months
  To evaluate postural balance used the variables: maximum displacement of the center of pressure, speed of displacement of the center of pressure and ground reaction forces as an impulse and braking

SECONDARY OUTCOMES:
Pain assessment during application of ice and shortwave diathermy | We evaluated 22 volunteers in a period of one year and 6 months
  To evaluate the pain during the application of the studied features we use the McGill questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Thiago B Muniz, Master, Principal Investigator — University of Sao Paulo
Locations (1):
- Rehabilitation Center HCRP, FMRP-USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Algafly AA, George KP. The effect of cryotherapy on nerve conduction velocity, pain threshold and pain tolerance. Br J Sports Med. 2007 Jun;41(6):365-9; discussion 369. doi: 10.1136/bjsm.2006.031237. Epub 2007 Jan 15. PMID 17224445
- [Background] Arsenault AB, Belanger AY, Durand MJ, De Serres SJ, Fortin L, Kemp F. Effects of TENS and topical skin anesthesia on soleus H-reflex and the concomitant influence of skin/muscle temperature. Arch Phys Med Rehabil. 1993 Jan;74(1):48-53. PMID 8420520
- [Background] Beaulieu M, Allard P, Simoneau M, Dalleau G, Hazime FA, Rivard CH. Relationship between oscillations about the vertical axis and center of pressure displacements in single and double leg upright stance. Am J Phys Med Rehabil. 2010 Oct;89(10):809-16. doi: 10.1097/PHM.0b013e3181f1b4af. PMID 20855981
- [Background] Beck TW, Housh TJ, Mielke M, Cramer JT, Weir JP, Malek MH, Johnson GO. The influence of electrode placement over the innervation zone on electromyographic amplitude and mean power frequency versus isokinetic torque relationships. J Neurosci Methods. 2007 May 15;162(1-2):72-83. doi: 10.1016/j.jneumeth.2006.12.009. Epub 2006 Dec 28. PMID 17275093
- [Background] Belaid D, Rougier P, Lamotte D, Cantaloube S, Duchamp J, Dierick F. [Clinical and posturographic comparison of patients with recent total hip arthroplasty]. Rev Chir Orthop Reparatrice Appar Mot. 2007 Apr;93(2):171-80. doi: 10.1016/s0035-1040(07)90221-4. French. PMID 17401291
- [Background] Bleakley CM, O'Connor S, Tully MA, Rocke LG, Macauley DC, McDonough SM. The PRICE study (Protection Rest Ice Compression Elevation): design of a randomised controlled trial comparing standard versus cryokinetic ice applications in the management of acute ankle sprain [ISRCTN13903946]. BMC Musculoskelet Disord. 2007 Dec 19;8:125. doi: 10.1186/1471-2474-8-125. PMID 18093299
- [Background] Bolgla LA, Uhl TL. Reliability of electromyographic normalization methods for evaluating the hip musculature. J Electromyogr Kinesiol. 2007 Feb;17(1):102-11. doi: 10.1016/j.jelekin.2005.11.007. Epub 2006 Jan 19. PMID 16423539
- [Background] Collins JJ, De Luca CJ. Open-loop and closed-loop control of posture: a random-walk analysis of center-of-pressure trajectories. Exp Brain Res. 1993;95(2):308-18. doi: 10.1007/BF00229788. PMID 8224055
- [Background] Deal DN, Tipton J, Rosencrance E, Curl WW, Smith TL. Ice reduces edema. A study of microvascular permeability in rats. J Bone Joint Surg Am. 2002 Sep;84(9):1573-8. PMID 12208913
- [Background] Dewhurst S, Macaluso A, Gizzi L, Felici F, Farina D, De Vito G. Effects of altered muscle temperature on neuromuscular properties in young and older women. Eur J Appl Physiol. 2010 Feb;108(3):451-8. doi: 10.1007/s00421-009-1245-9. Epub 2009 Oct 15. PMID 19830450
- [Background] Dewhurst S, Riches PE, De Vito G. Moderate alterations in lower limbs muscle temperature do not affect postural stability during quiet standing in both young and older women. J Electromyogr Kinesiol. 2007 Jun;17(3):292-8. doi: 10.1016/j.jelekin.2006.03.002. Epub 2006 May 15. PMID 16698285
- [Background] Farina D, Merletti R, Enoka RM. The extraction of neural strategies from the surface EMG. J Appl Physiol (1985). 2004 Apr;96(4):1486-95. doi: 10.1152/japplphysiol.01070.2003. PMID 15016793
- [Background] Faryniarz DA, Bhargava M, Lajam C, Attia ET, Hannafin JA. Quantitation of estrogen receptors and relaxin binding in human anterior cruciate ligament fibroblasts. In Vitro Cell Dev Biol Anim. 2006 Jul-Aug;42(7):176-81. doi: 10.1290/0512089.1. PMID 16948498
- [Background] Guirro RR, Forti F, Bigaton DR. Proposal for electrical insulation of the electromyographic signal acquisition module. Electromyogr Clin Neurophysiol. 2006 Nov;46(6):355-63. PMID 17147078
- [Background] Janwantanakul P. The effect of quantity of ice and size of contact area on ice pack/skin interface temperature. Physiotherapy. 2009 Jun;95(2):120-5. doi: 10.1016/j.physio.2009.01.004. Epub 2009 Mar 21. PMID 19627693
- [Background] Kernozek TW, Greany JF, Anderson DR, Van Heel D, Youngdahl RL, Benesh BG, Durall CJ. The effect of immersion cryotherapy on medial-lateral postural sway variability in individuals with a lateral ankle sprain. Physiother Res Int. 2008 Jun;13(2):107-18. doi: 10.1002/pri.393. PMID 18229881
- [Background] Kurca E, Drobny M. Four quantitative EMG methods and theirs individual parameter diagnostic value. Electromyogr Clin Neurophysiol. 2000 Dec;40(8):451-8. PMID 11155536
- [Background] Li S, Kukulka CG, Rogers MW, Brunt D, Bishop M. Sural nerve evoked responses in human hip and ankle muscles while standing. Neurosci Lett. 2004 Jul 1;364(2):59-62. doi: 10.1016/j.neulet.2004.01.084. PMID 15196677
- [Background] Lu G, Brittain JS, Holland P, Yianni J, Green AL, Stein JF, Aziz TZ, Wang S. Removing ECG noise from surface EMG signals using adaptive filtering. Neurosci Lett. 2009 Oct 2;462(1):14-9. doi: 10.1016/j.neulet.2009.06.063. Epub 2009 Jun 25. PMID 19559751
- [Background] Melnyk M, Faist M, Claes L, Friemert B. Therapeutic cooling: no effect on hamstring reflexes and knee stability. Med Sci Sports Exerc. 2006 Jul;38(7):1329-34. doi: 10.1249/01.mss.0000227635.86285.3b. PMID 16826031
- [Background] Norcross MF, Blackburn JT, Goerger BM. Reliability and interpretation of single leg stance and maximum voluntary isometric contraction methods of electromyography normalization. J Electromyogr Kinesiol. 2010 Jun;20(3):420-5. doi: 10.1016/j.jelekin.2009.08.003. Epub 2009 Sep 9. PMID 19744866
- [Background] Piedrahita H, Oksa J, Rintamaki H, Malm C. Effect of local leg cooling on upper limb trajectories and muscle function and whole body dynamic balance. Eur J Appl Physiol. 2009 Feb;105(3):429-38. doi: 10.1007/s00421-008-0920-6. Epub 2008 Nov 12. PMID 19002706
- [Background] Seigle B, Ramdani S, Bernard PL. Dynamical structure of center of pressure fluctuations in elderly people. Gait Posture. 2009 Aug;30(2):223-6. doi: 10.1016/j.gaitpost.2009.05.005. Epub 2009 Jun 2. PMID 19493680
- [Background] Vuillerme N, Sporbert C, Pinsault N. Postural adaptation to unilateral hip muscle fatigue during human bipedal standing. Gait Posture. 2009 Jul;30(1):122-5. doi: 10.1016/j.gaitpost.2009.03.004. Epub 2009 Apr 28. PMID 19403311
- [Background] Rattanachaiyanont M, Kuptniratsaikul V. No additional benefit of shortwave diathermy over exercise program for knee osteoarthritis in peri-/post-menopausal women: an equivalence trial. Osteoarthritis Cartilage. 2008 Jul;16(7):823-8. doi: 10.1016/j.joca.2007.10.013. Epub 2008 Feb 21. PMID 18178111
- [Background] Saeki Y. Effect of local application of cold or heat for relief of pricking pain. Nurs Health Sci. 2002 Sep;4(3):97-105. doi: 10.1046/j.1442-2018.2002.00112.x. PMID 12153407
- [Background] Rutkove SB, Kothari MJ, Shefner JM. Nerve, muscle, and neuromuscular junction electrophysiology at high temperature. Muscle Nerve. 1997 Apr;20(4):431-6. doi: 10.1002/(sici)1097-4598(199704)20:43.0.co;2-b. PMID 9121500
- [Background] Kiernan MC, Cikurel K, Bostock H. Effects of temperature on the excitability properties of human motor axons. Brain. 2001 Apr;124(Pt 4):816-25. doi: 10.1093/brain/124.4.816. PMID 11287380
- [Background] Dioszeghy P, Stalberg E. Changes in motor and sensory nerve conduction parameters with temperature in normal and diseased nerve. Electroencephalogr Clin Neurophysiol. 1992 Aug;85(4):229-35. doi: 10.1016/0168-5597(92)90110-w. PMID 1380909
- [Background] Garrett CL, Draper DO, Knight KL. Heat distribution in the lower leg from pulsed short-wave diathermy and ultrasound treatments. J Athl Train. 2000 Jan;35(1):50-5. PMID 16558608
- [Background] Nurse MA, Nigg BM. The effect of changes in foot sensation on plantar pressure and muscle activity. Clin Biomech (Bristol). 2001 Nov;16(9):719-27. doi: 10.1016/s0268-0033(01)00090-0. PMID 11714548
- [Derived] Muniz TB, Moraes R, Guirro RR. Lower limb ice application alters ground reaction force during gait initiation. Braz J Phys Ther. 2015 Mar-Apr;19(2):114-21. doi: 10.1590/bjpt-rbf.2014.0080. Epub 2015 Apr 27. PMID 25993625